CLINICAL TRIAL: NCT05568888
Title: A Prospective, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Large Simple Trial Evaluating the Use of BE1116 (4-Factor Prothrombin Complex Concentrate [Kcentra® / Beriplex®]) to Improve Survival in Patients With Traumatic Injury and Acute Major Bleeding
Brief Title: Evaluation of BE1116 in Patients With Traumatic Injury and Acute Major Bleeding to Improve Survival ( TAP Study )
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated early because mortality was lower than expected and a significant increase in sample size would have been required to meet statistical goals of the study. No safety reasons were involved in the decision to terminate the study.
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BE1116_3006; 2021-005060-21 (EudraCT Number)
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Injury
MeSH Terms: conditions — Wounds and Injuries | interventions — factor IX, factor VII, factor X, prothrombin drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BE1116 (Experimental): Administration by IV infusion
  Interventions: Drug: BE1116
- Placebo (Placebo Comparator): Administration by IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BE1116 — 4-Factor Prothrombin Complex administered by intravenous (IV) infusion
  Other Names: 4-Factor Prothrombin Complex; Kcentra®; Beriplex®
  Arms: BE1116
Drug: Placebo — Administered by IV infusion
  Arms: Placebo

SUMMARY:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled, parallel-group, large simple trial to investigate the efficacy and safety of a single intravenous (IV) infusion of BE1116 in subjects who have traumatic injury, with confirmed or suspected acute major bleeding and / or predicted to receive a large volume blood product transfusion.

ELIGIBILITY:
Inclusion Criteria:

* (a) Estimated age ≥ 15 years. Older minimum age is required in some locations. FOR United Kingdom: Estimated or actual age ≥ 16 years FOR Australia: Estimated or actual age ≥ 18 years AND (b) Estimated or actual weight ≥ 50 kg (110 lbs).
* Traumatic injury with confirmed or suspected acute major bleeding and/or Revised Assessment of Bleeding and Transfusion (RABT) score ≥ 2
* Activation of massive transfusion protocol

Exclusion Criteria:

* Healthcare professional cardiopulmonary resuscitation including chest compressions for ≥ 5 consecutive minutes at any time before randomization
* Isolated penetrating or blunt cranial injury, or exposed brain matter
* Isolated burns estimated to be > 20% total body surface area or suspected inhalational injury
* Known anticoagulation treatment or a history of a TEE, within the past 3 months.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1366 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (113):
- United States (90):
  - UAB Hospital, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - Chandler Regional Medical Center, Chandler, Arizona
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - Valleywise Medical Center, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - University Medical Center Tucson, Tucson, Arizona
  - UAMS Medical Center, Little Rock, Arkansas
  - LAC+USC Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Riverside University Health System Medical Center, Moreno Valley, California
  - UC Irvine, Orange, California
  - UC Davis Medical Center, Sacramento, California
  - UC San Diego Medical Center, San Diego, California
  - San Francisco General Hospital and Trauma Center, San Francisco, California
  - University of Colorado Aurora, Aurora, Colorado
  - UC Health Memorial Hospital Central, Colorado Springs, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Medical Center, Washington D.C., District of Columbia
  - George Washington University Hospital, Washington D.C., District of Columbia
  - UF Health Jacksonville, Jacksonville, Florida
  - University of Miami/Ryder Trauma Center, Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northeast Georgia Health System, Gainesville, Georgia
  - Atrium Health - Medical Center of central Georgia, Macon, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Methodist Hospital, Indianapolis, Indiana
  - St. Vincent's Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Kentucky Albert B. Chandler Hospital, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - University Medical Center of New Orleans, New Orleans, Louisiana
  - LSU Health Shreveport, Shreveport, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - University Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Hospital, Robbinsdale, Minnesota
  - Health Partners Regions Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center (UMMC), Jackson, Mississippi
  - SSM Health St. Louis, St Louis, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - UNMC (University of Nebraska Medical Center), Omaha, Nebraska
  - Cooper Health Care, Camden, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Capital Health Regional Medical Center, Trenton, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - NYU Langone, Mineola, New York
  - Jamaica Hospital Medical Center, Richmond Hill, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Mercy Health - St. Vincent Medical Center, Toledo, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - Oregon Health and Sciences University Hospital, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Presbyterian, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Brown University (Rhode Island Hospital), Providence, Rhode Island
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Erlanger Baroness Hospital, Chattanooga, Tennessee
  - University of Tennessee Medical Center - UTMCK, Knoxville, Tennessee
  - Regional Medical Center, Memphis, Tennessee
  - Vanderbilt Hospital and Clinics, Nashville, Tennessee
  - Dell Seton Medical Center, Austin, Texas
  - University Medical Center El Paso, El Paso, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - JPS Health Network (John Peter Smith Hospital), Fort Worth, Texas
  - Ben Taub General Hospital - Baylor Medical Center - Harris Health Network, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - University Hospital, San Antonio, Texas
  - UT Health Tyler, Tyler, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Harborview Medical Center, Seattle, Washington
  - J.W. Ruby Memorial Hospital, Morgantown, West Virginia
  - University Hospital, Madison, Wisconsin
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Australia (9):
  - Liverpool Hospital, Sydney, Liverpool
  - John Hunter Hospital, Sydney, New Lambton
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal Adelaide, Adelaide, South Australia
  - St. George Hospital, Kogarah, Sydney
  - Westmead Hospital, Westmead, Sydney
  - Royal Hobart Hospital, Hobart, Tasmania
  - Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- United Kingdom (14):
  - Queen Elizabeth Hospital, Birmingham
  - Southmead Hospital, Bristol
  - Cambridge Addenbrookes University, Cambridge
  - University Hospital Coventry, Coventry
  - Hull Royal Infirmary Hull University Teaching Hospitals NHS Trust, Hull
  - Leeds Teaching Hospital, Leeds
  - Aintree University Hospital, Liverpool
  - St. Georges Hospital, London
  - Imperial College Healthcare, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Queen's Medical Centre, Nottingham University Hospitals NHS Trust, Nottingham
  - John Radcliffe Hospital, Oxford
  - Sheffield Teaching Hospital, Sheffield
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 28 Mar 2023 to 29 October 2024 .
Pre-assignment Details: A total of 1366 participants were enrolled in this study. Of these, 1245 participants were treated as per their assigned treatment, either BE1116 or placebo.
Groups:
- BE1116: Participants received a single administration of BE1116 via intravenous (IV) administration on Day 1.
- Placebo: Participants received IV administration of placebo matched to BE1116.
Period: Overall Study
Arm/Group | BE1116 | Placebo
Started | 689 | 677
Treated | 618 | 627
Completed | 628 | 605
Not Completed | 61 | 72
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Deviation | 2 | 1
Not completed — Withdrawal by Subject/Legally Authorized Representative | 47 | 53
Not completed — Withdrawal by Parent/Guardian | 10 | 14
Not completed — No IP Administered/Subject Excluded | 1 | 4

BASELINE CHARACTERISTICS:
Population: Analysis was performed on Intent-to-treat (ITT) population, which included all randomized participants. In this population, analyses were based on the treatment to which participants were randomized, regardless of any treatment they received.
Groups:
- BE1116: Participants received a single administration of BE1116 via IV administration on Day 1.
- Total: Total of all reporting groups
Arm/Group | BE1116 | Placebo | Total
Number analyzed (Participants) | 689 | 677 | 1366
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (17.00) | 39.8 (17.65) | 40.2 (17.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 141 | 304
  Male | 526 | 536 | 1062
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 97 | 87 | 184
  Not Hispanic or Latino | 490 | 493 | 983
  Unknown or Not Reported | 102 | 97 | 199
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 12 | 21
  Asian | 13 | 21 | 34
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 201 | 210 | 411
  White | 350 | 335 | 685
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 108 | 93 | 201

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With All-cause 6-hour Mortality
Description: Here, the percentage of participants with all-cause mortality has been reported. Percentages were rounded off if the second digit after the decimal point is equal to or more than five.
Time Frame: Up to 6 hours after randomization
Population: Analysis was performed on the ITT and modified ITT (mITT) population. The ITT population included all the randomized participants. The mITT population included all participants from ITT population who received at least one complete or partial dose of the investigational product (IP) (BE1116 or placebo). It also included participants with a missing or non-testable Glasgow Coma Score, or a score less than 15, as well as those who received blood product transfusions prior to randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | BE1116 | Placebo
Number analyzed (Participants) | 689 | 677
Percentage of participants
  All-cause Mortality in ITT Analysis Set | 7.3 | 4.6
  All-cause Mortality in mITT Analysis Set: number analyzed (Participants) | 432 | 436
  All-cause Mortality in mITT Analysis Set | 7.2 | 4.1
Statistical Analysis 1: Comparison: BE1116 vs Placebo; Null hypotheses: The all-cause 6-hour mortality rates in BE1116 is no better than the control; Test type: Superiority — A Bayesian logistic regression model was used to compare all-cause 6-hour mortality rate between the BE1116 and placebo arms. The null hypothesis is rejected if the posterior probability of 6-hour mortality rate difference (BE1116-placebo) being negative is greater than predefined threshold at interim and final analyses (ITT population); p = 1.9, Regression, Logistic — Reported value reflect a posterior probability difference rather than p-value; Estimated difference Placebo - BE1116 = -2.5, 95% CI 2-sided [-5.02 to -0.13] — Reported values reflect a 95% Credible Interval rather than a 95% Confidence Interval
Statistical Analysis 2: Comparison: BE1116 vs Placebo; Null hypotheses: The all-cause 6-hour mortality rates in BE1116 is no better than the control; Test type: Superiority — A Bayesian logistic regression model was used to compare all-cause 6-hour mortality rate between the BE1116 and placebo arms. The null hypothesis is rejected if the posterior probability of 6-hour mortality rate difference (BE1116-placebo) being negative is greater than predefined threshold at interim and final analyses (mITT population); p = 3.1, Regression, Logistic — Reported value reflect a posterior probability difference rather than p-value; Estimated difference Placebo - BE1116 = -2.8, 95% CI 2-sided [-5.80 to 0.13] — Reported values reflect a 95% Credible Interval rather than a 95% Confidence Interval

2. Secondary Outcome: Proportion of Participants With All-cause 24-hour In-hospital Mortality
Description: In-hospital mortality up to 24 hours after randomization was recorded and assessed for the primary hospitalization only. Here, the percentage of participants with all-cause in hospital mortality has been reported. Percentages were rounded off if the second digit after the decimal point is equal to or more than five.
Time Frame: Up to 24 hours after randomization
Population: As planned, analysis was performed on the mITT population. The mITT population included all participants from ITT population who received at least one complete or partial dose of BE1116 or placebo. It also included participants with a missing or non-testable Glasgow Coma Score, or a score less than 15, as well as those who received blood product transfusions prior to randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | BE1116 | Placebo
Number analyzed (Participants) | 432 | 436
Percentage of participants | 11.1 | 7.3
Statistical Analysis 1: Comparison: BE1116 vs Placebo; Null hypotheses: The all-cause 24-hour in-hospital mortality rates in BE1116 is no better than the control; Test type: Superiority — A Bayesian logistic regression model was used to compare all-cause 24-hour in-hospital mortality rate between the BE1116 and placebo arms. The null hypothesis is rejected if the posterior probability of 24-hour in-hospital mortality rate difference (BE1116-placebo) being negative is greater than predefined threshold at interim and final analyses (mITT population); p = 3.0, Regression, Logistic — Reported value reflect a posterior probability difference rather than p-value; Estimated difference Placebo - BE1116 = -3.6, 95% CI 2-sided [-7.35 to 0.15] — Reported values reflect a 95% Credible Interval rather than a 95% Confidence Interval

3. Secondary Outcome: Proportion of Participants With All-cause In-hospital Mortality Up to 30 Days After Randomization
Description: In-hospital mortality was recorded and assessed for the primary hospitalization only. Here, the percentage of participants with all-cause in hospital mortality has been reported. Percentages were rounded off if the second digit after the decimal point is equal to or more than five.
Time Frame: Up to 30 days after randomization
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | BE1116 | Placebo
Number analyzed (Participants) | 432 | 436
Percentage of participants | 24.8 | 18.6
Statistical Analysis 1: Comparison: BE1116 vs Placebo; Null hypotheses: The all-cause 30 days in-hospital mortality rates in BE1116 is no better than the control; Test type: Superiority — A Bayesian logistic regression model was used to compare all-cause 30 days in-hospital mortality rate between the BE1116 and placebo arms. The null hypothesis is rejected if the posterior probability of 30 days in-hospital mortality rate difference (BE1116-placebo) being negative is greater than predefined threshold at interim and final analyses (mITT population); p = 1.4, Regression, Logistic — Reported value reflect a posterior probability difference rather than p-value; Estimated difference Placebo - BE1116 = -6.0, 95% CI 2-sided [-11.42 to -0.68] — Reported values reflect a 95% Credible Interval rather than a 95% Confidence Interval

4. Secondary Outcome: Proportion of Participants Who Underwent Surgical or Interventional Radiological Procedures to Stop Bleeding Related to the Primary Injury
Description: Here, the percentage of participants with who underwent surgical or interventional radiological procedures to stop bleeding related to the primary injury has been reported. Percentages were rounded off if the second digit after the decimal point is equal to or more than five.
Time Frame: Up to 24 hours after randomization
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | BE1116 | Placebo
Number analyzed (Participants) | 432 | 436
Percentage of participants | 78.0 | 75.5
Statistical Analysis 1: Comparison: BE1116 vs Placebo; Null hypotheses: The proportion of subjects who undergo surgical or interventional radiological procedures to stop bleeding related to the primary injury up to 24 hours in BE1116 is no better than the control; Test type: Superiority — A Bayesian logistic regression model was used to compare difference in proportion of subjects between the BE1116 and placebo arms. The null hypothesis is rejected if the posterior probability of subjects who undergo surgical or interventional radiological procedures to stop bleeding related to the primary injury up to 24 hours difference (BE1116-placebo) being negative is greater than predefined threshold at interim and final analyses (mITT population); p = 18.9, Regression, Logistic — Reported value reflect a posterior probability difference rather than p-value; Estimated difference Placebo - BE1116 = -2.5, 95% CI 2-sided [-7.98 to 3.05]; Reported values reflect a 95% Credible Interval rather than a 95% Confidence Interval

5. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (SAEs)
Description: The number of participants with treatment-emergent SAEs considered related to IP that occurred during primary hospitalization within the 30 days after randomization are summarized by treatment arm.
Time Frame: Up to 30 days after randomization
Population: Analysis was performed on the safety population. The safety population included of all the participants from ITT population who received at least one complete or partial dose of BE1116 or placebo, based on the treatment actually received.
Measure: Number; unit: Count of participants
Arm/Group | BE1116 | Placebo
Number analyzed (Participants) | 618 | 627
Count of participants | 34 | 46

6. Secondary Outcome: Number of Participants With In-hospital Overall and Related Thromboembolic Events (TEEs)
Description: The TEEs may be symptomatic or asymptomatic, and arterial or venous (eg, deep vein thrombosis, pulmonary embolism, ischemic stroke [including thromboembolic stroke], myocardial infarction). The observed in-hospital overall and related to IP TEEs are reported here.
Time Frame: Up to 30 days after randomization
Population: as for outcome 5
Measure: Number; unit: Count of participants
Arm/Group | BE1116 | Placebo
Number analyzed (Participants) | 618 | 627
Count of participants
  Overall TEEs | 133 | 139
  Related TEEs | 46 | 51

7. Secondary Outcome: Number of Participants With Acute Respiratory Distress Syndrome (ARDS)
Description: ARDS will be assessed using the Berlin definition based on four criteria: timing, chest imaging, origin of edema, oxygenation (mild, moderate or severe) and high-flow nasal oxygen.
Time Frame: Up to 30 days after randomization
Population: as for outcome 5
Measure: Number; unit: Count of participants
Arm/Group | BE1116 | Placebo
Number analyzed (Participants) | 618 | 627
Count of participants | 31 | 28

8. Secondary Outcome: Number of Participants With Multiple Organ Failure
Description: Multiple organ failure will be assessed using the Denver post injury multiple organ failure score. The Denver score rates the dysfunction of 4 organ systems (pulmonary, renal, hepatic, and cardiac), which are each graded on a scale from 0 to 3, where 0 represents "mild" and 3 was "severe". Multiple organ failure is defined as a score > 3.
Time Frame: Up to 30 days after randomization
Population: as for outcome 5
Measure: Number; unit: Count of participants
Arm/Group | BE1116 | Placebo
Number analyzed (Participants) | 618 | 627
Count of participants | 59 | 53

9. Secondary Outcome: Number of Participants With Acute Kidney Injury (AKI) Requiring Renal Replacement Therapy
Description: Renal replacement therapy included dialysis, hemofiltration, or hemodiafiltration. AKI according to the Kidney Disease Improving Global Outcomes (KDIGO) guidelines is diagnosed if any one of the following happens: • Serum creatinine increases by ≥ 0.3 mg/dL (≥ 26.5 μmol/L) within 48 hours • Serum creatinine increases to ≥ 1.5 times the baseline level, within the past 7 days • Urine levels drops to less than 0.5 mL/kg/hour for 6 hours
Time Frame: Up to 30 days after randomization
Population: as for outcome 5
Measure: Number; unit: Count of participants
Arm/Group | BE1116 | Placebo
Number analyzed (Participants) | 618 | 627
Count of participants | 52 | 29

ADVERSE EVENTS:
Time Frame: Up to 30 days after randomization
Description: The safety analysis (analyses of serious adverse events (SAEs) and non-serious adverse events) is based on the Safety Population, which included all participants who received at least one complete or partial dose of BE1116 or placebo. All-cause mortality data were analyzed using the ITT population, comprising all randomized participants, classified according to their randomized treatment assignments.
Arm/Group | BE1116 | Placebo
All-Cause Mortality (participants affected / at risk) | 146/689 | 114/677
Serious Adverse Events (participants affected / at risk) | 203/618 | 168/627
Other Adverse Events (participants affected / at risk) | 32/618 | 39/627
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BE1116 (N=618) | Placebo (N=627)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 42 (44) | 48 (50)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 21 (21)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 5 (5)
Acute Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 50 (50) | 24 (24)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal infarct (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 30 (32) | 21 (21)
Peripheral artery thrombosis (Vascular disorders) | 4 (5) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 2 (2) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 2 (3) | 5 (5)
Shock (Vascular disorders) | 2 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 2 (2)
Peripheral vein occlusion (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 6 (6)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 25 (25) | 27 (28)
Septic shock (Infections and infestations) | 8 (8) | 8 (8)
Sepsis (Infections and infestations) | 5 (6) | 5 (6)
Abdominal abscess (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Empyema (Infections and infestations) | 2 (2) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
Necrotising soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Retroperitoneal abscess (Infections and infestations) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 2 (2)
Liver abscess (Infections and infestations) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 43 (44) | 36 (36)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Dehiscence (General disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 6 (6) | 3 (3)
Cerebral infarction (Nervous system disorders) | 3 (3) | 3 (3)
Embolic stroke (Nervous system disorders) | 2 (2) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 2 (2) | 2 (2)
Parietal lobe stroke (Nervous system disorders) | 2 (2) | 0 (0)
Carotid artery thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Diplegia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2)
Middle cerebral artery stroke (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 2 (2)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Paroxysmal sympathetic hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
Spinal epidural haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 8 (9) | 7 (8)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Failure to anastomose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fat embolism (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post transfusion purpura (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pancreatic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ureteric injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abdominal wall wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 1 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Procedural pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic necrosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Acute cholecystitis necrotic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Perforation bile duct (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pelvic fluid collection (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Antithrombin III deficiency (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BE1116 (N=618) | Placebo (N=627)
Deep vein thrombosis (Vascular disorders) | 32 (41) | 39 (44)

LIMITATIONS AND CAVEATS:
The study was terminated due to feasibility reasons. No safety issues contributed to the decision to terminate the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT05568888/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT05568888/SAP_001.pdf